CLINICAL TRIAL: NCT02719158
Title: A 1-Month, Prospective, Multicenter, Randomized, Dose-Ranging, Sham-Controlled, Blinded Study of OTO-201 Given as a Single Administration for Treatment of Acute Otitis Media With Tympanostomy Tubes in Pediatric Subjects
Brief Title: Dose Ranging Study of OTO-201 in AOMT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otonomy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201-201508
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Results first posted 2020-09-24 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Acute Otitis Media; AOMT
Keywords: Acute otitis media with tympanostomy tubes; OTIPRIO
MeSH Terms: conditions — Otitis Media | interventions — Ciprofloxacin; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- 6 mg OTO-201 (Experimental): 6 mg OTO-201 (sustained-release suspension of ciprofloxacin), single 0.1 mL supra-tympanostomy tube (STT) administration to the affected ear(s)
  Interventions: Drug: 6 mg ciprofloxacin
- 12 mg OTO-201 (Experimental): 12 mg OTO-201 (sustained-release suspension of ciprofloxacin), single 0.2 mL supra-tympanostomy tube (STT) administration to the affected ear(s)
  Interventions: Drug: 12 mg ciprofloxacin
- Sham (empty syringe) (Sham Comparator): Sham (empty syringe), single 0.1 mL STT administration to the affected ear(s)
  Interventions: Other: Sham

INTERVENTIONS:
Drug: 6 mg ciprofloxacin — Single administration of OTO-201
  Other Names: OTIPRIO
  Arms: 6 mg OTO-201
Drug: 12 mg ciprofloxacin — Single administration of OTO-201
  Other Names: OTIPRIO
  Arms: 12 mg OTO-201
Other: Sham
  Arms: Sham (empty syringe)

SUMMARY:
Dose Ranging Study of OTO-201 in AOMT

DETAILED DESCRIPTION:
This is a 1-month, prospective, multicenter, randomized, dose-ranging, sham-controlled, blinded study in which eligible subjects with either unilateral or bilateral acute otitis media with tympanostomy tubes (AOMT) will receive a single administration of 6 mg OTO-201, 12 mg OTO-201, or sham into the affected ear(s).

ELIGIBILITY:
Inclusion Criteria includes, but is not limited to:

* Subject is a male or female aged 6 months to 17 years, inclusive
* Subject has a clinical diagnosis of acute otitis media with tympanostomy tubes (AOMT)
* Subject's caregiver is willing to comply with the protocol an attend all study visits

Exclusion Criteria includes, but is not limited to:

* Subject has a history of sensorineural hearing loss
* Subject has tympanic membrane perforation other than the surgical tympanostomy tube perforation
* Subject has a history of known immunodeficiency disease

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl LeBel, PhD, Study Chair — Otonomy, Inc.
Locations (1):
- Contact Otonomy call center for trial locations, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Sham Control: simulated, single administration
Period: Overall Study
Arm/Group | 6 mg OTO-201 | 12 mg OTO-201 | Control
Started | 38 | 38 | 19
Completed | 38 | 38 | 18
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: 95 subjects randomized (19 sham, 38 6mg, 3812mg OTO-201). 1 sham and 1 6mg subject positive for Group A strep and not in intento to treat (ITT) population (Baseline and efficacy) leaving 18 sham, 37-6mg OTO-201, 38-12 mg OTO-201 in ITT. Safety population (AE/SAE) = randomized (19 sham, 38 6mg, 38 12mg).
Groups:
- Total: Total of all reporting groups
Arm/Group | 6 mg OTO-201 | 12 mg OTO-201 | Control | Total
Number analyzed (Participants) | 37 | 38 | 18 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.004 (3.0546) | 3.955 (2.9111) | 3.551 (2.4583) | 3.498 (2.8915)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 7 | 40
  Male | 22 | 20 | 11 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 2 | 8
  Not Hispanic or Latino | 33 | 35 | 16 | 84
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 9 | 5 | 22
  White | 29 | 27 | 11 | 67
  More than one race | 0 | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 37 | 38 | 18 | 93

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events
Description: Number of subjects with adverse events during the study from dosing up to 1 month after dosing
Time Frame: Up to 1 month
Population: Safety analysis set: all subjects who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 6 mg OTO-201 | 12 mg OTO-201 | Control
Number analyzed (Participants) | 38 | 38 | 19
Participants | 19 | 14 | 4

2. Primary Outcome: Otoscopic Examination: Auricle and Meatus
Description: Number of affected ears (i.e., those ears that were infected) whose external ear and ear canal (auricle and meatus), when examined through an otoscope, appeared normal at Baseline and appeared abnormal at Day 29. The auricle and meatus of each infected ear was examined using an otoscope and was assessed as either normal or abnormal at every visit. This outcome looks to see if there was a worsening of the condition of the auricle and meatus with treatment (i.e., a safety measure).
Time Frame: Up to 1 month
Population: Safety Population (19 sham, 38 6mg, 38 12 mg) who could have had one or 2 affected ears at Baseline (that is, it was not necessary for both ears to be infected to take part in the study). This is why the number of ears in each group do not equal twice the number of participants.
Measure: Number; unit: abnormal affected ears at Day 29
Units Other Than Participants: normal affected ears at Baseline
Arm/Group | 6 mg OTO-201 | 12 mg OTO-201 | Control
Number analyzed (Participants) | 38 | 38 | 19
Number analyzed (normal affected ears at Baseline) | 21 | 17 | 7
abnormal affected ears at Day 29 | 2 | 0 | 0

3. Primary Outcome: Otoscopic Examination: Tympanic Membrane
Description: Number of affected ears (i.e., those ears that were infected) whose ear drum (tympanic membrane), when examined through an otoscope, appeared normal at Baseline and appeared abnormal at Day 29. The tympanic membrane of each infected ear was examined using an otoscope and was assessed as either normal or abnormal at every visit. This outcome looks to see if there was a worsening of the condition of the tympanic membrane with treatment (i.e., a safety measure).
Time Frame: Up to 1 month
Population: as for outcome 2
Measure: Number; unit: abnormal ears at Day 29
Units Other Than Participants: normal affected ears at Baseline
Arm/Group | 6 mg OTO-201 | 12 mg OTO-201 | Control
Number analyzed (Participants) | 38 | 38 | 19
Number analyzed (normal affected ears at Baseline) | 23 | 15 | 10
abnormal ears at Day 29 | 1 | 0 | 0

4. Secondary Outcome: Absence of Otorrhea
Description: Absence of otorrhea (middle ear drainage)
Time Frame: Up to Two Weeks
Population: Modified intent-to-treat analysis set: all subjects who were randomized, received treatment, did not have group A streptococci cultured on Visit 1 (Day 1), and had at least 1 on-therapy visit.
Measure: Count of Participants; unit: Participants
Arm/Group | 6 mg OTO-201 | 12 mg OTO-201 | Control
Number analyzed (Participants) | 37 | 38 | 18
Participants | 20 | 23 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were reported during dosing and up to 1 month following dosing.
Arm/Group | 6 mg OTO-201 | 12 mg OTO-201 | Control
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38 | 0/19
Other Adverse Events (participants affected / at risk) | 5/38 | 6/38 | 1/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 6 mg OTO-201 (N=38) | 12 mg OTO-201 (N=38) | Control (N=19)
Otitis media acute (Infections and infestations) | 4 | 1 | 1
Pyrexia (General disorders) | 1 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication subject to Sponsor consent.